CLINICAL TRIAL: NCT04966442
Title: GrandAides; a Workforce Innovation to Address Post Acute Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Temple University
Record Dates: First submitted 2021-06-07; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GrandAides (Experimental): Patients randomized to this arm of the trial received access to a specially trained GrandAide to work as a credible messenger community health worker. This GrandAide received 6 weeks of education around congestive heart failure to support the patient in the outpatient setting.
  Interventions: Behavioral: GrandAides
- Standard of Care (No Intervention): This arm served as the control and included standard of care outpatient support for patients with heart failure.This support was done telephonically.

INTERVENTIONS:
Behavioral: GrandAides — Enhanced post acute care for patients recently admitted for congestive heart failure
  Arms: GrandAides

SUMMARY:
Randomized controlled trial with two groups looking at post hospital care for patients who were admitted with congestive heart failure. The control group includes standard of care provided to the patients after discharge including a hospital employed community health worker. The intervention group receives a specially trained GrandAide following the GrandAide model for post acute care. Difference in ER visits and readmissions was measured.

DETAILED DESCRIPTION:
GrandAides program is a credible messenger community health worker based program that assumes a community health worker from the community who has specialized education around a certain chronic condition will be able to support patients in the outpatient setting more effectively than current standard of care. In this study a GrandAide visited a patient discharged from the hospital in their home for 4 weeks providing education, checking vital signs, and assisting with communication with the cardiologist. The study measured the difference in hospital admissions and ER visits between the group that was assigned a GrandAid and the group that took part in standard care. The groups were assigned randomly. The difference was calculated using one and two tailed t-test results.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of heart failure Lives in 6 zipcode catchment area of Temple University Hospital Is followed by Temple Cardiology

Exclusion Criteria:

End Stage Renal Disease Housed in a Skilled Nursing Facility Substance Use Disorder Unable to give consent Doesn't speak English Under age 18

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
ER visits | 3 years
  number of ER visits

IPD SHARING:
Plan to Share IPD: Undecided